CLINICAL TRIAL: NCT05871775
Title: Effects of Therapeutic Intervention Through Selective Functional Movement Assessment on Pain, Function, Balance and Gait in Patients With Chronic Nonspecific Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Hyun-Joong Kim, investigator, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21040966ABN012212HSR2822
Record Dates: First submitted 2023-04-24; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Chronic Nonspecific Neck Pain
Keywords: exercise; neck pain; chronic pain
MeSH Terms: conditions — Motor Activity; Neck Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized exercise (Experimental)
  Interventions: Behavioral: Personalized exercise
- Stabilization exercise (Active Comparator)
  Interventions: Behavioral: Stabilization exercise
- General exercise (Active Comparator)
  Interventions: Behavioral: General exercise

INTERVENTIONS:
Behavioral: Personalized exercise — After selective functional movement evaluation, customized interventions for each patient
  Arms: Personalized exercise
Behavioral: Stabilization exercise — Neck stabilization exercise and sensorimotor program
  Arms: Stabilization exercise
Behavioral: General exercise — General mobility exercise and strength exercise program
  Arms: General exercise

SUMMARY:
According to the order of the physical examination, the scope of the problem is narrowed down by excluding the parts of the body that do not have problems and adjusting the load related to stability. A list of problems can be created through an algorithmic approach that guesses which structures will have problems through active or passive movement. This provides an optional therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 65 who have experienced chronic neck pain for more than 12 weeks (Blanpied et al., 2017).
* Those with more than moderate pain (4/10 cm) on the visual analogue scale (VAS) (Paksaichol et al., 2012).
* Those with a neck disability index (NDI) of mild disability (5/50 score) or higher (Lluch et al., 2014).
* Those who consented to participate in this study.

Exclusion Criteria:

* Patients with severe pathology such as radiation pain due to intervertebral disc herniation or neurological signs consistent with tumor, whiplash injury, cervical vertebra fracture, or nerve root compression.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
neck disability index | change from baseline neck disability index at 8weeks
  The questionnaire was composed of 10 questions to provide information on how neck pain affects daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Dajeong Kim, MSc, Principal Investigator — Yongin University
Locations (1):
- Yongin University, Yŏngin, South Korea

IPD SHARING:
Plan to Share IPD: No
Only information provided in the paper publication is included.